CLINICAL TRIAL: NCT00143936
Title: The Safety and Efficacy of Low and High Carbohydrate Diets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Gary D. Foster, PhD, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT001103 (NIH); 1R01AT001103-01 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Obesity
Keywords: Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Carb (Active Comparator): Low Cabohydrate Diet: 20 week of weekly group behavior modification, 20 weekly bi-weekly, bi-monthly to finish
  Interventions: Behavioral: Low- Carbohydrate -Atkins Diet
- Low Calorie (Active Comparator): Low Calorie Diet: 20 weeks of weekly behavior modification, 20 weekly of bi-weekly, bimonthly to finish 2 years
  Interventions: Behavioral: Low Calorie Diet

INTERVENTIONS:
Behavioral: Low- Carbohydrate -Atkins Diet — Low Carbohydrate Diet
  Other Names: low carb
  Arms: Low Carb
Behavioral: Low Calorie Diet — Maintain a low calorie diet
  Other Names: low cal
  Arms: Low Calorie

SUMMARY:
This study will compare the safety and effectiveness of a low carbohydrate diet (Atkins Diet) with a high carbohydrate diet (conventional USDA diet).

DETAILED DESCRIPTION:
Despite the considerable mass appeal of popular diet books, such diet approaches lack data to support their efficacy and safety. Despite its widespread use for more than 30 years, the Atkins diet has never been evaluated in a large, randomized, controlled trial. This study will assess the short-term and long-term clinical effects of a low-carbohydrate diet and a high-carbohydrate diet in overweight and obese men and women.

Participants in this study will be randomly assigned to the Atkins diet (low-carbohydrate, unlimited fat and protein) or a conventional USDA diet (high-carbohydrate, low fat). The study will evaluate the effects of each dietary approach on changes in: 1) weight and body composition, 2) metabolic and organ function, 3) exercise tolerance. Each participant will be enrolled in the study for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 30 and 40
* Live and work within 1 hour of the study site
* Stable psychological status

Exclusion Criteria:

* History of heart disease, heart attack, or stroke
* Blood pressure > 140/90 mmHG
* Abnormal cholesterol levels
* Significant psychiatric illness
* Any medication that affects weight or metabolic rate
* Presence or history of a chronic disease that is known to affect appettite, food intake, or metabolism (i.e. diabetes, thyroid disease or cancer).
* Currently using antidepressants, steroids, tobacco or illegal drugs
* Pregnant, breastfeeding, or planning pregnancy
* 10 lb change in weight within 6 months of study entry
* History of malignant arrhythmias or cerebrovascular, renal, or hepatic disease
* History of protein wasting diseases or gout
* Severe arthritis
* Osteoperosis
* Certain types of hormone replacement therapy
* Currently following a vegetarian diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foster, PhD, Principal Investigator — University of Pennsylvania; Holly Wyatt, MD, Principal Investigator — University of Colorado, Denver; James Hill, PhD, Principal Investigator — University of Colorado, Denver; Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Washington University, St Louis, Missouri
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Friedman AN, Ogden LG, Foster GD, Klein S, Stein R, Miller B, Hill JO, Brill C, Bailer B, Rosenbaum DR, Wyatt HR. Comparative effects of low-carbohydrate high-protein versus low-fat diets on the kidney. Clin J Am Soc Nephrol. 2012 Jul;7(7):1103-11. doi: 10.2215/CJN.11741111. Epub 2012 May 31. PMID 22653255
- [Derived] Borradaile KE, Halpern SD, Wyatt HR, Klein S, Hill JO, Bailer B, Brill C, Stein RI, Miller BV 3rd, Foster GD. Relationship between treatment preference and weight loss in the context of a randomized controlled trial. Obesity (Silver Spring). 2012 Jun;20(6):1218-22. doi: 10.1038/oby.2011.216. Epub 2011 Jul 14. PMID 21760633
- [Derived] Foster GD, Wyatt HR, Hill JO, Makris AP, Rosenbaum DL, Brill C, Stein RI, Mohammed BS, Miller B, Rader DJ, Zemel B, Wadden TA, Tenhave T, Newcomb CW, Klein S. Weight and metabolic outcomes after 2 years on a low-carbohydrate versus low-fat diet: a randomized trial. Ann Intern Med. 2010 Aug 3;153(3):147-57. doi: 10.7326/0003-4819-153-3-201008030-00005. PMID 20679559